CLINICAL TRIAL: NCT03943771
Title: Effect on Pre-operative Anxiety of a Personalized Three-dimensional Kidney Model Prior to Nephron-sparing Surgery for Renal Tumor.
Acronym: R3DP-A
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Schedule issue
Sponsor: University Hospital, Bordeaux (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: CHUBX 2017/58
Record Dates: First submitted 2019-05-07; First posted 2019-05-09 (Actual); Last update posted 2020-01-27 (Actual); Status verified 2020-01

CONDITIONS: Kidney Neoplasms; Carcinoma, Renal Cell
Keywords: Kidney Neoplasms; Carcinoma, Renal Cell; Nephron-Sparing Surgery; 3D Modeling; 3D Printing; Anxiety; Personalized Medicine
MeSH Terms: conditions — Kidney Neoplasms; Carcinoma, Renal Cell; Anxiety Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Virtual modelization group (Experimental): Patients having their kidney modelized in three dimensions on a software
  Interventions: Other: Anxiety, renal anatomy and surgery questionnaires
- Printed modelization group (Experimental): Patients having their kidney modelized and printed in three dimensions
  Interventions: Other: Anxiety, renal anatomy and surgery questionnaires
- Control group (Sham Comparator): No kidney model
  Interventions: Other: Anxiety, renal anatomy and surgery questionnaires

INTERVENTIONS:
Other: Anxiety, renal anatomy and surgery questionnaires — The day before surgery, all the patients will be visited by a member of the investigator team for preoperative consultation and will be given a questionnaire evaluating their anxiety based on STAI and VAS scores. The two experimental groups will be offered their renal modelization to be manipulated (virtually or physically) before the questionnaire.
  A second survey assessing basic renal anatomy and surgery understanding will also be completed by the patients.
  Anxiolytics prescription prior to surgery will be collected inside the medical file.

SUMMARY:
Investigators aimed to estimate the effect of showing and handling a three-dimensional modelization of a patient's kidney presenting with tumor the day before his nephron-sparing surgery. The main outcome measure was the effect on anxiety assessed via the STAI score. 2 types kidney models (virtual and printed) will be evaluated as compared to usual information, using a randomization.

DETAILED DESCRIPTION:
Announcement of serious illnesses and especially cancerous diseases has major impacts on one's psychological field. Need of surgery can create even other fears due to its unknown nature. Use of tools to decrease anxiety and enhance understanding prior to surgery is a key point in comprehensive care that is way not enough promoted for now. In the field of surgery, available methods to deal with pre-operative anxiety are massively represented by anxiolytics drugs, only few other devices were evaluated.

Technological development in healthcare has seen the rising of three-dimensional media, especially in surgery, for procedure planning. There is no doubt that this tool is effective in helping surgeons regarding the studies published within the past few years but there is no such evidence concerning the benefit for patients. Some authors report improvement of patients understanding and great satisfaction referring to the usefulness of this tool. But none of these papers evaluated anxiety.

The goal of our research is to measure the effect of a personalized three-dimensional model of patients' kidney on pre-operative anxiety.

For this purpose investigators will randomly assign a total of 66 patients planned to have a nephron-sparing surgery for kidney tumor in 3 different groups. Inside the 2 interventional groups, patients' kidneys will be modelized in three dimensions, one group will then be 3D-printed.

The third group will be control with usual preoperative information. The day before surgery, 3D models will be presented to their respective owner. All patients will have to complete a survey evaluating their anxiety level and also their understanding of renal anatomy and surgical procedure.

ELIGIBILITY:
Inclusion Criteria:

* Consecutive patients presenting with renal tumor allowing a nephron-sparing surgery
* Participating in UroCCR database
* Having a contrast abdominal scanner prior to surgery
* Owing social insurance contract
* Inpatient surgery

Exclusion Criteria:

* Unable to give informed consent
* No contrast scanner

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2019-07 (Estimated); Primary Completion 2020-04 (Estimated); Study Completion 2020-04 (Estimated)

PRIMARY OUTCOMES:
State-anxiety score of the State-Trait Anxiety Inventory (STAI) questionnaire | The day before renal surgery, up to 1 month after inclusion
  Min : 20 = few anxiety Max : 80 = severe anxiety
Visual Analog Scale (VAS) score for anxiety | The day before renal surgery, up to 1 month after inclusion
  Min : 0 = no anxiety Max : 10 = maximum anxiety

SECONDARY OUTCOMES:
Renal anatomy and surgical strategies questionnaire score | The day before renal surgery, up to 1 month after inclusion
  Renal anatomy : min/max = 0/13, higher values represent a better understanding Surgical strategies : min/max = 0/7, higher values represent a better understanding
Anxiolytics prescription before surgery | The day before renal surgery, up to 1 month after inclusion
Pain numeric scale score | The day after renal surgery, up to 1 month after inclusion
  Min : 0 = no pain Max : 10 = maximum pain

CONTACTS AND LOCATIONS:
Locations (1):
- CHU de Bordeaux, Bordeaux, France